CLINICAL TRIAL: NCT01998737
Title: Point-of-care Osteoporosis Diagnostics With Bindex® Pocket Size Instrument and FRAX
Status: Completed | Type: Observational
Sponsor: Bone Index Finland Ltd (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Bind03; BoneIndex03 (Other: Bone Index Finland Ltd.)
Record Dates: First submitted 2013-11-25; First posted 2013-12-02 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Osteoporosis
Keywords: Osteoporosis, diagnostics, ultrasound
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Women under osteoporosis suspicion
- Healthy women

SUMMARY:
Osteoporosis is a disease that leads to impaired skeletal strength and increased fracture risk. Among 200 million osteoporotic patients (Tarantino, Cannata et al. 2007) most are diagnosed only after several fractures. Furthermore, the progressively aging population will increase the prevalence of osteoporosis. It is estimated that over 75% of osteoporotic patients are not diagnosed and does not receive treatment for their condition.

In this study we aim to investigate the strength of Density Index (DI) for prediction of proximal femur and lumbar spine BMD as well as determining the diagnostic thresholds for DI for osteoporosis diagnostics by using the International Society for Clinical Densitometry guidelines. In addition we aim to investigate how many additional women would be identified for osteoporosis diagnosis/ treatment based on adding FRAX to Bindex versus adding FRAX to DXA.

The investigators will start and organize a multicenter study in 5 osteoporosis clinics in Suomen Terveystalo Healthcare Service Company in Finland. A total of 1100 postmenopausal women (age 50 -79 years) will be measured with both axial DXA and Bindex. In addition, the FRAX questioinnaire will be asked from everybody attending the study.

Clinical hypotheses:

1. Cortical bone thickness is decreased in osteoporosis.
2. Patient age, weight and height are related to BMD status and therefore are needed in BMD estimation (Density Index).
3. Ultrasound is a safe method in osteoporosis screening and diagnostics for osteoporosis.
4. Fracture risk factors (FRAX) and point-of-care bone density measurement together have significantly higher sensitivity and specificity for osteoporosis/treatment decisions than one method alone.

DETAILED DESCRIPTION:
The following procedures will be applied

* Signing Informed Consent
* Filling in the FRAX questionnaire
* DXA measurements of the proximal femur and AP spine
* Bindex ultrasound measurement of both the tibia and the radius

Written informed consent is obtained from all subjects before enrolment to the study. All patient data is coded, i.e. made anonymous, to conform to personal data protection. The data is processed only for study purposes.

A total of 1100 postmenopausal women (age 50 -79 years) will participate the study. The subjects will be divided into two groups: healthy (100 women) and under osteoporosis suspicion (1000 women). The groups will be matched by BMI.

Written informed consent is obtained from all subjects before enrolment in the study. All patient data is coded, i.e. made anonymous, to conform to personal data protection. The data is processed only for study purposes.

ELIGIBILITY:
Osteoporosis suspicion

Inclusion Criteria:

* Age: 50 - 59 years (n = 500) and 60-79 years (n = 500).
* Post-menopausal status.
* At least one of the clinical risk factors for fracture:

  * Low body mass index (< 19kg/m2)
  * Previous fragility fracture
  * Parental history of hip fracture
  * Glucocorticoid treatment (≥ 5mg prednisolone daily or equivalent for 3 months or more)
  * Current smoking
* Alcohol intake 3 or more units daily
* Causes of secondary osteoporosis:

  * Untreated hypogonadism
  * Inflammatory bowel disease
  * Prolonged immobility
  * Organ transplantation
  * Type 1 and type 2 diabetes
  * Thyroid disorders
  * Chronic obstructive pulmonary disease
* A Physician has referred the woman to axial DXA investigation.

Exclusion Criteria:

* Treatment: osteoporosis medication.
* Obesity: body mass index BMI > 30kg/m2
* a refusal to participate in the study

Healthy

Inclusion Criteria:

* Age: 50 - 59 years (n = 50) and 60-79 years (n = 50).
* Post-menopausal status.
* No diseases or treatments which may affect to bone health.

Exclusion Criteria:

* Treatment: osteoporosis medication.
* a refusal to participate in the study
* Obesity: body mass index BMI > 30kg/m2

Ages: 50 Years to 79 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 1100 postmenopausal women (age 50 -79 years) will participate the study. The subjects will be divided into two groups: healthy (100 women) and under osteoporosis suspicion (1000 women). The groups will be matched by BMI.
  Women for the under osteoporosis suspicion group will be invited from those who have got a referral for DXA examination from their doctor.
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heikki Kröger, MD, PhD, Principal Investigator — Kuopio University Hospital; Janne P Karjalainen, PhD, Study Director — Bone Index Finland Ltd; Ossi Riekkinen, PhD, Study Director — Bone Index Finland Ltd
Locations (6):
- Finland (6):
  - Terveystalo Kamppi, Helsinki
  - Terveystalo Jyväskylä, Jyväskylä
  - Terveystalo Kouvola, Kouvola
  - Kuopio University Hospital, Kuopio
  - Terveystalo Lahti, Lahti
  - Terveystalo Mikkeli Marski, Mikkeli

RESULTS

PARTICIPANT FLOW:
Groups:
- Women Under Osteoporosis Suspicion: Subjects with at least one risk factor for osteoporotic fracture.
- Healthy Women: In healthy group females without risk factors for fracture or diseases affecting bone health were recruited.
Period: Overall Study
Arm/Group | Women Under Osteoporosis Suspicion | Healthy Women
Started | 911 | 100
Completed | 888 | 100
Not Completed | 23 | 0
Not completed — Corrupted database | 23 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Women Under Osteoporosis Suspicion | Healthy Women | Total
Number analyzed (Participants) | 888 | 100 | 988
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 453 | 74 | 527
  >=65 years | 435 | 26 | 461
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (7) | 61.6 (6.6) | 64.9 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 888 | 100 | 988
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 888 | 100 | 988
Region of Enrollment [Number; unit: participants]
  Finland | 888 | 100 | 988
Weight [Mean (Standard Deviation); unit: kg] | 64.2 (9.9) | 65.5 (9.2) | 64.4 (9.9)
Height [Mean (Standard Deviation); unit: cm] | 161.5 (6.1) | 162.3 (6.1) | 161.5 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of the Density Index Against Dual Energy X-ray Absorptiometry for Detecting Osteoporosis
Description: The thresholds for the Density Index (DI) in osteoporosis diagnostics in comparison to dual energy x-ray absorptiometry (DXA) are evaluated in independent population.
Time Frame: 3 years
Measure: Number; unit: percentage of true positives
Groups:
- Women Under Osteoporosis Suspicion; Healthy Women: As defined in the protocol
Arm/Group | Women Under Osteoporosis Suspicion | Healthy Women
Number analyzed (Participants) | 888 | 100
percentage of true positives | 93.7 | 100

2. Primary Outcome: Specificity of the Density Index Against Dual Energy X-ray Absorptiometry for Detecting Osteoporosis
Description: as for outcome 1
Time Frame: 3 years
Measure: Number; unit: percentage of true negatives
Arm/Group | Women Under Osteoporosis Suspicion | Healthy Women
Number analyzed (Participants) | 888 | 100
percentage of true negatives | 81.6 | 93.8

3. Secondary Outcome: Number of Participants That Would Require Additional DXA Examination to Confirm Diagnosis
Description: The previously determined thresholds have been applied. The results show amount of subject whose DI value is between the thresholds. These subjects would need DXA measurement to verify diagnosis.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Women Under Osteoporosis Suspicion | Healthy Women
Number analyzed (Participants) | 888 | 100
Participants | 288 | 27

ADVERSE EVENTS:
Time Frame: Study duration 3 years
Arm/Group | Women Under Osteoporosis Suspicion | Healthy Women
Serious Adverse Events (participants affected / at risk) | 0/888 | 0/100
Other Adverse Events (participants affected / at risk) | 0/888 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No